CLINICAL TRIAL: NCT00004314
Title: Phase II Pilot Study of Aminoimidazole Carboxamide Riboside (AICAR), a Precursor of Purine Synthesis, for Lesch-Nyhan Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, San Diego (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11823; UCSD-733
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Lesch-Nyhan Syndrome
Keywords: Lesch-Nyhan syndrome; inborn errors of metabolism; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Lesch-Nyhan Syndrome; Metabolism, Inborn Errors; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Drug: aminomidazole carboxamide riboside

SUMMARY:
OBJECTIVES: I. Determine the effects of aminoimidazole carboxamide riboside (AICAR) on hematologic manifestations of Lesch-Nyhan disease.

II. Assess the behavioral and neurological benefits of AICAR in patients with Lesch-Nyhan disease.

III. Examine the effect of AICAR on purine production.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

After a 3-day baseline, patients are treated with aminoimidazole carboxamide riboside (AICAR) by continuous infusion for 12 days. Concurrent allopurinol and folate are allowed.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Men with Lesch-Nyhan syndrome Moderate erythrocyte macrocytosis No active urinary tract disease or impaired renal function

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2
Dates: Start 1996-02

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barshop, Study Chair — University of California, San Diego

REFERENCES:
- [Background] Page T, Barshop BA, Yu A, et al.: Treatment of Lesch-Nyhan syndrome with AICAR. In: Sahota A, Tayor M, eds.: Purine and Pyrimidine Metabolism in Man VIII. Plenum Press, New York, NY: 1995, pp 353-356.
- [Background] Page T, Barshop B, Yu AL, Nyhan WL. Treatment of Lesch-Nyhan syndrome with AICAR. Adv Exp Med Biol. 1994;370:353-6. doi: 10.1007/978-1-4615-2584-4_76. No abstract available. PMID 7660927